CLINICAL TRIAL: NCT03840018
Title: Randomized Trial to Assess the Effectiveness of a Postal Intervention for Reducing the Chronic Use of Highe Doses of Proton Pump Inhibitors
Brief Title: Effectiveness of a Postal Intervention to Improve the Use of PPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osakidetza (Other)
Responsible Party: Principal Investigator, Elena Valverde, Primary care pharmacist, Osakidetza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EVB-IBP-2017-01
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Drug Overdose
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Sending doctors the lists of patients that meet the inclusion criteria to have their treatment reviewed
- Letter by post to patients (Other): Patients were sent a letter explaining the risks of using PPIs at long-term high doses and encouraging them to visit their doctor
  Interventions: Other: Letter by post to patients

INTERVENTIONS:
Other: Letter by post to patients — Patients received an informative letter by post, in which their doctor invited them to seek an appointment for a medication review
  Arms: Letter by post to patients

SUMMARY:
It was a randomised intervention study, with before-and-after outcome measures and a control group, in patients who had an active long-term prescription for PPIs at high doses for at least 6 months.

DETAILED DESCRIPTION:
The intervention consisted of sending patients an informative letter by post, in which their doctor invited them to seek an appointment for a medication review. Control group patients did not receive such a letter, and they were treated as usual (their doctors received a list of identifiers of patients on high doses).

The main outcome variable was the number of active prescriptions of each PPI dose (high dose/standard dose/treatment cessation) at 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the care of our organisation who in May 2017 had an active long-term prescription for PPIs at high doses for at least 6 months.

Exclusion Criteria:

* Patients whose GPs declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Active prescriptions of each proton pump inhibitors dose after the intervention | 6 months
  Number of active prescriptions of each proton pump inhibitors dose (high dose/standard dose/treatment cessation) at 6 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elena Valverde, Principal Investigator — Osakidetza
Locations (1):
- Bidasoa Integrated Health Organization, Hondarribia, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: No